CLINICAL TRIAL: NCT01279785
Title: A Phase 1 Pilot Study of 123I-MIP-1072 Single Photon Emission Computed Tomography (SPECT)/CT Imaging With Optional Compact Gamma Camera Probe Imaging in Men With Prostate Cancer Undergoing Prostatectomy
Brief Title: A Pilot Study of 123I-MIP-1072 SPECT/CT Imaging With Optional Compact Gamma Camera Probe Imaging in Men With Prostate Cancer Undergoing Prostatectomy
Status: Withdrawn | Type: Observational
Why Stopped: Similar study to be completd once kit for new formulation becomes available.
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TX-P104
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
Keywords: Molecular Imaging; PSMA; adenocarcinoma; prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate Cancer Patients: Male participants who are scheduled to undergo standard of care prostatectomy for presumed localized prostate cancer at the NIH Clinical Center and have evidence of a recent (within 12 months of study entry) trans-rectal biopsy documenting adenocarcinoma of the prostate.
  Interventions: Drug: 123I-MIP-1072

INTERVENTIONS:
Drug: 123I-MIP-1072 — Single IV dose
  Other Names: Trofex

SUMMARY:
This is a single arm, open label study of up to 20 patients with prostate cancer scheduled for prostatectomy at the NIH Clinical Center. 123I-MIP-1072 image data will be evaluated for visible uptake and compared with histopathology.

DETAILED DESCRIPTION:
This is an exploratory, single arm, open label pilot study evaluation of 123I-MIP-1072 intraprostatic uptake determination by SPECT/CT imaging (and optional CGCP imaging), with histological confirmation of disease localization and staging. Methodical evaluation of 123I-MIP-1072 in intraprostatic tumorous and non-tumours regions will provide important preliminary data upon which further clinical studies can be based. The optional additional CGCP imaging was added, because of its inherent potential for higher resolution scintigraphic detection of 123I-MIP-1072 localization. This imaging feasibility data will provide important preliminary information for the use of CGCP imaging in prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be scheduled to undergo standard of care prostatectomy for presumed localized prostate cancer at the NIH Clinical Center.
* Have had or will undergo multiparametric endorectal coil 3T MR at the NIH clinical center
* Recent (within 12 months of study entry) trans-rectal biopsy indicating the presence of adenocarcinoma of the prostate gland
* Participant must be 18 years or older.
* ECOG Performance grade of 0 to 2. (see Appendix 1)
* Ability to understand and provide informed consent. All subjects must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.
* Participants of childbearing potential must agree to use an acceptable form of birth control, defined as abstinence, barrier or other acceptable, effective contraceptive method until 7 days after the infusion of study drug.

Exclusion Criteria:

* Participants for whom participating would significantly delay the scheduled standard of care therapy.
* Subjects must not have prostate biopsies performed within 12 weeks before imaging; or within 8 weeks before imaging providing that the absence of hemorrhage is confirmed by MR imaging.
* SGOT and SGPT ≥ 2 x of the upper limits of normal; total bilirubin, of ≥ 1.5 x the upper limits of normal or ≥ 3.0 mg/dl in patients with Gilbert's syndrome.
* Administered a radioisotope within 5 physical half lives prior to study enrollment.
* Patients with severe claustrophobia unresponsive to oral anxiolytics
* Subjects weighing ≥350 lbs or are unable to fit within the imaging gantry
* Subjects who have received androgen deprivation therapy.
* Subjects with any medical condition or other circumstances that, in the opinion of the Investigator, would significantly decrease obtaining reliable data, achieving study objectives or completing the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to twenty adult men with biopsy confirmed prostate cancer scheduled for prostatectomy at the NIH Clinical Center will undergo 123I-MIP-1072 SPECT/CT and optional CGCP imaging prior to prostatectomy. These patients will also have undergone/will undergo multi-parametric 3T MR imaging at NIH which is considered standard of care at NIH clinical center.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the tissue distribution of 123I-MIP-1072 SPEC/CT imaging in tumor and non-tumorous regions of the prostate (as determined by histopathology) in patients undergoing standard of care prostatectomy | Evaulated through Day 30

SECONDARY OUTCOMES:
To evaluate the potential of 123I-MIP-1072 imaging to predict malignancy as defined by histopathology and multiparametric 3T MR | Evaulated through Day 30
To further evaluate the safety of 123I-MIP-1072 | Evaluated through Day 30
To evaluate the intensity of 123I-MIP-1072 uptake with respect to Gleason Grade | Evaluated through Day 30
To evaluate the intensity of 123I-MIP-1072 uptake with respect to PSMA expression | Evaluated through Day 30
To evaluate feasibility of imaging123I-MIP-1072 uptake using an FDA-approved compact endorectal gamma camera probe (CGCP) | Evaluated through Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Peter Choyke, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- CCR/NCI - Molecular Imaging Program, Bethesda, Maryland, United States